CLINICAL TRIAL: NCT04322162
Title: Addressing Sleep Apnea Post-Stroke (ASAP)
Brief Title: Addressing Sleep Apnea Post-Stroke/TIA
Acronym: ASAP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: IIR 16-211; 1I01HX002324-01A2 (NIH)
Record Dates: First submitted 2020-03-24; First posted 2020-03-26 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Ischemic Stroke; Transient Ischemic Attack (TIA); Obstructive Sleep Apnea
Keywords: Ischemic stroke; Transient ischemic attack (TIA); Stepped-wedge trial; Implementation Science; Hybrid Type I; Quality Improvement; Systems Redesign; Champion; External Facilitation; Audit and feedback; Local Adaptation; Obstructive Sleep Apnea; Polysomnography; Sustainability; Business-case
MeSH Terms: conditions — Ischemic Stroke; Ischemic Attack, Transient; Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Active implementation - Wave 1 (First and Second Sites) (Experimental): This four-year stepped-wedge evaluation includes a total of 6 sites. Active implementation is initiated in 3 waves, each of which includes 2 sites. The project involves two phases at each of the 6 sites: a variable number of 7-month data periods during baseline period (three 7-month periods for Wave 1 sites, four 7-month data periods for Wave 2 sites, five 7-month data periods for Wave 3 sites), three 7-month data periods in active implementation phase for each wave. Wave 1 and Wave 2 sites will also each have one 7-month period of sustainability. The stepped-wedge design allows for 6 mutually exclusive, 7-month data periods. The baseline data period is the time prior to the date of the baseline site visit. The active implementation data period extends 21 months after the site visit. The stepped-wedge design allows site-level estimates of proportions on six different cross-sectional samples. Investigators will have repeated information on each site. "Arm" 1 corresponds to Wave 1.
  Interventions: Other: ASAP Intervention Quality Improvement Protocol
- Active implementation - Wave 2 (Third and Fourth Sites) (Experimental): This four-year stepped-wedge evaluation includes a total of 6 sites. Active implementation is initiated in 3 waves, each of which includes 2 sites. The project involves two phases at each of the 6 sites: a variable number of 7-month data periods during baseline period (three 7-month periods for Wave 1 sites, four 7-month data periods for Wave 2 sites, five 7-month data periods for Wave 3 sites), three 7-month data periods in active implementation phase for each wave. Wave 1 and Wave 2 sites will also each have one 7-month period of sustainability. The stepped-wedge design allows for 6 mutually exclusive, 7-month data periods. The baseline data period is the time prior to the date of the baseline site visit. The active implementation data period extends 21 months after the site visit. The stepped-wedge design allows site-level estimates of proportions on six different cross-sectional samples. Investigators will have repeated information on each site. "Arm" 2 corresponds to Wave 2.
  Interventions: Other: ASAP Intervention Quality Improvement Protocol
- Active implementation - Wave 3 (Fifth and Sixth Sites) (Experimental): This four-year stepped-wedge evaluation includes a total of 6 sites. Active implementation is initiated in 3 waves, each of which includes 2 sites. The project involves two phases at each of the 6 sites: a variable number of 7-month data periods during baseline period (three 7-month periods for Wave 1 sites, four 7-month data periods for Wave 2 sites, five 7-month data periods for Wave 3 sites), three 7-month data periods in active implementation phase for each wave. Wave 1 and Wave 2 sites will also each have one 7-month period of sustainability. The stepped-wedge design allows for 6 mutually exclusive, 7-month data periods. The baseline data period is the time prior to the date of the baseline site visit. The active implementation data period extends 21 months after the site visit. The stepped-wedge design allows site-level estimates of proportions on six different cross-sectional samples. Investigators will have repeated information on each site. "Arm" 3 corresponds to Wave 3.
  Interventions: Other: ASAP Intervention Quality Improvement Protocol

INTERVENTIONS:
Other: ASAP Intervention Quality Improvement Protocol — The intervention program includes: (1) a systems redesign Virtual Collaborative, and; (2) data monitoring and is designed to aid each of the 6 participating VAMCs in developing, implementing, and evaluating the implementation of an acute OSA testing and treatment protocol for ischemic stroke/TIA patients. The sites will choose a diagnostic strategy (i.e., unattended polysomnography [PSG]/home sleep test [HST], in-laboratory PSG, direct to auto-titrating [auto]-PAP) and a therapeutic strategy (i.e., in-laboratory PAP titration, auto-PAP). The intervention will employ 3 implementation strategies: (1) local adaptation; (2) external facilitation, and; (3) audit and feedback.

SUMMARY:
Effectively identifying and treating risk factors for ischemic stroke and transient ischemic attack (TIA) is important to patients, their family members, and healthcare systems. While obstructive sleep apnea (OSA) is a known risk factor for stroke and TIA that is present in more than 70% of stroke/TIA survivors, testing for OSA is infrequently performed for patients and within healthcare systems. The Addressing Sleep Apnea Post-Stroke/TIA (ASAP) study intends to improve rates of guideline-recommended OSA testing and treatment through local quality improvement initiatives (QI) conducted within and across 6 VA Medical Centers. ASAP will also determine the impact of these local QI initiatives on rates of OSA diagnosis, OSA treatment, recurrent vascular events, and hospital readmissions.

DETAILED DESCRIPTION:
Approximately 11,000 Veterans present to a VAMC annually with an acute ischemic stroke or TIA. The cornerstone of secondary stroke/TIA prevention includes delivering timely, guideline-concordant vascular risk factor management. Over the past decade, OSA has been recognized as a potent, underdiagnosed, and inadequately treated cerebrovascular risk factor. OSA is very common among patients with stroke/TIA with a prevalence of 60-80%. Despite being highly prevalent, 70-80% of patients with OSA are neither diagnosed nor treated. Untreated OSA has been associated with poor outcomes among patients with cerebrovascular disease including higher mortality and worse functional status. The mainstay of OSA therapy is positive airway pressure (PAP). PAP reduces recurrent vascular events, improves neurological symptoms and functional status among stroke/TIA patients with OSA. The evidence favoring neurological recovery is strongest when interventions are applied early post-stroke/TIA. Guidelines recommend diagnosing and treating OSA for stroke and TIA patients; however, within VHA, very few stroke or TIA patients receive OSA screening. This guideline recommendation was informed in part by clinical trials utilizing an acute OSA assessment protocol developed and implemented by the investigators' group. To address the observed gap in care, the investigators propose a Hybrid Type I, randomized, stepped-wedge trial at 6 VAMCs to increase the rate of timely, guideline-concordant diagnosis and treatment of OSA among Veterans with ischemic stroke/TIA and thereby reduce recurrent vascular events and hospital readmissions. The investigators will identify matched control sites for each ASAP implementation site to examine temporal trends in outcomes among non-intervention sites. For example, the investigators will use administrative data to examine the use of polysomnography across stroke/TIA patients in the VA system and compare changes in matched controls versus the intervention sites on the diagnostic rate. The same adjustment approach will be used for ASAP intervention sites and for control sites.

ELIGIBILITY:
Inclusion Criteria:

As recruitment was at the facility-level, an ASAP a VAMCS had to have >50 stroke/TIA admissions per year and have at least 1.0 FTE staff dedicated to systems redesign

* The sites were chosen because they are diverse in terms of geography and sleep infrastructure

  * Local site investigators and their care teams will identify patients eligible for the QI intervention, specifically patients with ischemic stroke/TIA without a prior diagnosis of OSA

Exclusion Criteria:

* VAMCs were excluded if they had <=50 stroke/TIA admissions per year and did not have at least 1.0 FTE staff dedicated to systems redesign
* Local site investigators and their care teams will prioritize the protection of patients from harm and use their clinical expertise in identifying patients who would not be candidates for PAP therapy

  * e.g., palliative care/hospice, inability to use PAP therapy [e.g., orofacial injury], or contraindication to PAP [e.g., inability to clear secretions]

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-04-02 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Facility-level OSA diagnostic rate | 30-day
  PSG completion or initiation of auto-PAP within 30 days of presentation for the index stroke or TIA

SECONDARY OUTCOMES:
Facility-level treatment rate | 30-day
  PAP initiation within 30 days of presentation to the facility. For this outcome, the denominator will be patients diagnosed with OSA. Patients with a prior diagnosis of sleep apnea and those who die within 7 days of presentation will be excluded. Because the denominator in this secondary effectiveness measure includes the patients who are diagnosed with OSA, it is variable and depends on the primary effectiveness outcome of diagnostic rate.
Facility-level recurrent vascular event rate | 90-day
  Stroke, myocardial infarction (MI), acute coronary syndrome (ACS), hospitalization for congestive heart failure (CHF), and all-cause mortality. The recurrent vascular event rate is measured from the day of presentation (e.g., to the Emergency Department) which may be the same as or prior to the day of admission.
Facility-level all-cause readmission rate | 90-day
  Includes an inpatient admission for any cause at either a VA or non-VA acute care facility.
Facility-level treatment rate (Positive airway pressure and non-positive airway pressure treatments) | 30-day
  PAP or non-PAP treatment initiation within 30 days of presentation to the facility. For this outcome, the denominator will be patients diagnosed with OSA. Patients with a prior diagnosis of sleep apnea and those who die within 7 days of presentation will be excluded. Because the denominator in this secondary effectiveness measure includes the patients who are diagnosed with OSA, it is variable and depends on the primary effectiveness outcome of diagnostic rate.

OTHER OUTCOMES:
Implementation Outcome - Adaptation | Measured throughout active implementation and sustainability periods
  Information regarding implementation of acute OSA diagnosis and treatment approaches will be collected at each site on an ongoing basis during brief phone calls every month between the local RA and/or local champion with members of the ASAP implementation team using the "local adaptation real-time tracking system" developed by a team of VA investigators. Local adaptations will also be recorded by local RAs in response to the monthly site assessments.
External Facilitation | Measured throughout active implementation and sustainability periods
  External facilitation changes over time based on the needs of the team. However, the core elements of relationship-building, methods training, communication, facilitating team-based problem solving, and monitoring performance over time will be preserved through external facilitation from a Lean Six Sigma Black belt experienced in stroke QI work and ASAP investigators experienced in implementation of post-stroke/TIA OSA programs. External facilitation activities will be recorded and will later be classified by type of contact, topic, and dose/duration.
Audit and Feedback | Measured throughout active implementation and sustainability periods
  To support the sites' use of data, the local teams will receive explicit training in team-based reflecting & evaluating, goal-setting, and planning. Meeting as a group, local teams will be encouraged to formally ask and answer questions like: "How are we doing?" "Are we where we want to be?" "What performance goals do we want to set as targets?" "What do we need to do to achieve our goals?" "How will we know how far or how close we are to hitting our targets?." Data usage will be monitored by the web-based data platform known as the ASAP "hub."
Sustainability - mixed methods analysis | Measured throughout sustainability period
  The sustainability analysis will include: a comparison of the change in the diagnostic rate from the baseline data period to the sustainability period. This will be obtained from the multilevel models as described for the Aim 1 analysis. The investigators will explore whether sites that use HST as their primary diagnostic approach, that continue to actively review their audit and feedback data, and that have champions who continue to engage with systems redesign demonstrate the greatest program sustainability.
Sustainability - Program Sustainability Assessment Tool (PSAT) | Measured prior to and at the end of active implementation period and at the end of the sustainability period
  Those agreeing to participate will receive a link to complete the Program Sustainability Assessment Tool (PSAT), an online tool which allows users to: (1) understand factors associated with sustainability; (2) assess the sustainability of a program; (3) review their sustainability report, and; (4) develop an action plan to enhance the chances of programmatic sustainability. This tool assesses the facility's overall capacity for sustainability and across the specific domains of: environmental support, funding stability, partnerships, organizational capacity, program adaptation, communications, and strategic planning. Reports are generated by this tool, ranking the facility from 1 (little to no extent) to 7 (to a great extent) and provides guidance on what areas can be addressed to maximize sustainability.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Jonathon Sico, MD MHS, Principal Investigator — VA Connecticut Healthcare System West Haven Campus, West Haven, CT; Dawn M. Bravata, MD, Principal Investigator — Richard L. Roudebush VA Medical Center, Indianapolis, IN
Locations (2):
- United States (2):
  - VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut
  - Richard L. Roudebush VA Medical Center, Indianapolis, IN, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Diaz MM, Hu X, Fenton BT, Kimuli I, Lee A, Lindsey H, Bigelow JK, Maiser S, Altalib HH, Sico JJ. Prevalence of and characteristics associated with in-hospital mortality in a Ugandan neurology ward. BMC Neurol. 2020 Jan 31;20(1):42. doi: 10.1186/s12883-020-1627-5. PMID 32005185
- [Result] Sico JJ, Sarwal A, Benish SM, Busis NA, Cohen BH, Das RR, Finsilver S, Halperin JJ, Kelly AG, Meunier L, Phipps MS, Thirumala PD, Villanueva R, von Gaudecker J, Bennett A, Shenoy AM. Quality improvement in neurology: Neurology Outcomes Quality Measurement Set. Neurology. 2020 Jun 2;94(22):982-990. doi: 10.1212/WNL.0000000000009525. Epub 2020 May 12. No abstract available. PMID 32398356
- [Result] Patel K, Nussbaum E, Sico J, Merchant N. Atypical case of Miller-Fisher syndrome presenting with severe dysphagia and weight loss. BMJ Case Rep. 2020 May 27;13(5):e234316. doi: 10.1136/bcr-2020-234316. PMID 32467120
- [Result] Arling G, Perkins A, Myers LJ, Sico JJ, Bravata DM. Blood Pressure Trajectories and Outcomes for Veterans Presenting at VA Medical Centers with a Stroke or Transient Ischemic Attack. Am J Med. 2022 Jul;135(7):889-896.e1. doi: 10.1016/j.amjmed.2022.02.012. Epub 2022 Mar 12. PMID 35292287
- [Result] Miech EJ, Perkins AJ, Zhang Y, Myers LJ, Sico JJ, Daggy J, Bravata DM. Pairing regression and configurational analysis in health services research: modelling outcomes in an observational cohort using a split-sample design. BMJ Open. 2022 Jun 7;12(6):e061469. doi: 10.1136/bmjopen-2022-061469. PMID 35672067
- [Result] Sico JJ, Koo BB, Perkins AJ, Burrone L, Sexson A, Myers LJ, Taylor S, Yarbrough WC, Daggy JK, Miech EJ, Bravata DM. Impact of the coronavirus disease-2019 pandemic on Veterans Health Administration Sleep Services. SAGE Open Med. 2023 May 3;11:20503121231169388. doi: 10.1177/20503121231169388. eCollection 2023. PMID 37152838
- [Result] Waddell KJ, Myers LJ, Perkins AJ, Sico JJ, Sexson A, Burrone L, Taylor S, Koo B, Daggy JK, Bravata DM. Development and validation of a model predicting mild stroke severity on admission using electronic health record data. J Stroke Cerebrovasc Dis. 2023 Sep;32(9):107255. doi: 10.1016/j.jstrokecerebrovasdis.2023.107255. Epub 2023 Jul 18. PMID 37473533
- [Derived] Bravata DM, Perkins AJ, Myers LJ, Daggy JK, Sexson A, Taylor SE, Burrone L, Koo BB, Miech EJ, Rattray N, Story KM, Waddell KJ, Ding QP, Sico JJ; ASAP Investigators Group. Quality Improvement Intervention to Increase Sleep Apnea Diagnostic Testing After Stroke and Transient Ischemic Attack: A Cluster Randomized Trial. JAMA Netw Open. 2025 Nov 3;8(11):e2543385. doi: 10.1001/jamanetworkopen.2025.43385. PMID 41236739
- [Derived] Bravata DM, Myers LJ, Perkins AJ, Sexson AE, Daggy JK, Taylor SE, Burrone L, Koo BB, Miech EJ, Rattray NA, Story KM, Waddell K, Ding Q, Sico JJ. Addressing sleep apnea post-stroke and transient ischemic attack (ASAP) clinical trial design features: Inclusion of usual care control sites and electronic health record data validation. Contemp Clin Trials. 2025 Dec;159:108135. doi: 10.1016/j.cct.2025.108135. Epub 2025 Oct 30. PMID 41173184